CLINICAL TRIAL: NCT03877536
Title: Antiretroviral Therapy for Acute HIV Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feeder cohort study closed.
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV 392; WRAIR 2393 (Other: WRAIR)
Record Dates: First submitted 2018-09-26; First posted 2019-03-15 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: prospective, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Genvoya 150Mg-150Mg-200Mg-10Mg Tablet (Experimental): Genvoya® (Elvitegravir, corbiscistat, Emtricitabine and Tenofovir Alafenamide): once a day antiretroviral pill starting within 1 week of enrollment.
  Interventions: Drug: Genvoya 150Mg-150Mg-200Mg-10Mg Tablet

INTERVENTIONS:
Drug: Genvoya 150Mg-150Mg-200Mg-10Mg Tablet — Participants will receive 1 tablet per day throughout study duration (96 weeks).

SUMMARY:
This study will evaluate the virologic effect, safety and tolerability of Genvoya® in adults during early acute HIV infection.

DETAILED DESCRIPTION:
This is a prospective, open-label study to describe the effects of early antiretroviral (ART) therapy on 1) viral load, 2) safety and tolerability of Genvoya®, 3) clinical outcomes and secondarily on HIV-specific immune responses. This study is a sub-study of RV 217 that will recruit participants with incident HIV diagnoses from the parent RV 217 cohort. Potential RV 392 volunteers will be recruited from the RV 217 ECHO cohort if they have been diagnosed with incident HIV Infection. Screening procedures for HIV in RV 217 are designed to identify participants during acute HIV infection (AHI) or early HIV infection. Participants will initiate Genvoya®, a once a day antiretroviral pill within 1 week of enrollment. RV 392 follow-up visits will largely overlap with RV 217 visits for the study duration of 96 weeks, but additional visits will occur early after initiation of Genvoya®. RV 392 participants will remain co-enrolled in RV 217 (i.e., RV 217 visits also continue); blood collection will be coordinated by the RV 392 team by prioritizing safety labs and then research labs within the allotted blood volumes while still meeting scientific objectives for both RV 217 and RV 392. Blood tests that are required for both protocols will only be collected once and will not be duplicated across the two protocols.

ELIGIBILITY:
Inclusion Criteria:

1. First identified as an incident HIV infection within one year of estimated time of infection in RV 217.
2. Willing to begin Genvoya® as soon as entering this study but not later than 7 days from study enrollment.
3. Successfully passed Test of Understanding (TOU) with a score of 80% or more on ten questions after three attempts.
4. Adult from 18 to 50 years of age.
5. Able to participate for 96 weeks of study visits
6. In general good health as determined by the PI or his/her designee
7. Willing to have photo or fingerprint taken for identification purposes
8. No history of ART for any reason, i.e., treatment naïve and no HIV-post-exposure prophylaxis (PEP) or HIV-pre-exposure prophylaxis (PrEP)) within 90 days prior to enrollment
9. Willing to have blood samples collected and stored.
10. Adequate renal function: estimated creatine clearance of >50 mL/min according to the Cockroft Gault formula 2 weeks prior to enrollment
11. Urine clean catch: glucose < trace and protein <1+ or as per site-specification 2 weeks prior to enrollment
12. Weight is > 35 kg
13. Female (only women of childbearing potential) Specific Criteria:

Negative pregnancy test 48 hours prior to enrollment:

Commits to continued use of adequate birth control method for 96 weeks of the study and prior to receiving study ART. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted, underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), condoms, diaphragms, intrauterine device (IUD), or abstinence. If depending on hormonal contraception, check package insert for drug interactions and/or consider adding a second barrier method.

Exclusion Criteria:

1. Any chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer, including but not limited to chronic hepatitis, renal insufficiency or failure; clinically significant forms of drug or alcohol abuse, mental illness, severe asthma, psychiatric disorders, heart disease, or cancer; or a physical finding on examination considered indicative of significant disease such as murmur (other than functional), hepatosplenomegaly, focal neurological deficit, etc.
2. Untreated AIDS-related opportunistic infection
3. An AIDS defining condition diagnosed within 30 days
4. Positive Hepatitis B surface antigen at any time in the past
5. Requiring use of any medication that is contraindicated with Genvoya®. See Appendix I and the package insert
6. Women who are breast-feeding

There are no inclusion/exclusion criteria based on CD4 count because CD4 count can be transiently diminished during acute HIV infection and ART initiation during early or acute HIV infection offers the potential benefit of limiting reservoir seeding and preventing immune destruction regardless of peripheral CD4 count at the time of treatment initiation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-17 (Estimated); Primary Completion 2023-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
Plasma viral load | Measured at 48 weeks after enrollment
  The number of study participants with plasma viral load <50 copies/mL
Plasma viral load | Measured at 96 weeks after enrollment
  The number of study participants with plasma viral load <50 copies/mL
Drug-related AEs and SAEs | Measured through week 96
  Occurrence of drug-related adverse events and serious adverse events at any time from enrollment up to 96 weeks after enrollment early HIV infection.
Treatment Discontinuation for AEs up to 96 weeks | Measured through week 96
  Tolerability of treatment as measured by treatment discontinuation for AEs up to 96 weeks

SECONDARY OUTCOMES:
CD4+ T cell count change | Measured over 48 weeks
  CD4+ T cell count change over first 48 weeks as compared to baseline.following the initiation of Genvoya®
Frequency of HIV-related illnesses | Measured through week 96
  Frequency of HIV-related illnesses (including acute retroviral syndrome)
Duration of HIV-related illnesses | Measured through week 96
  Duration of HIV-related illnesses (including acute retroviral syndrome)

OTHER OUTCOMES:
Changes in HIV-specific immune responses over time | Measured through week 96
  Description of changes in HIV-specific immune responses over time as characterized by intracellular cytokine staining (ICS)
Host humoral (IgG) responses | Measured through week 96
  Characterization of evolution in host humoral (IgG) responses to HIV envelope over time including development of neutralizing antibody responses
Markers of Immune Activation | Measured through week 96
  Description of markers of immune activation (soluble and cellular markers) by ICS.
HIV reservoir size | Measured through week 96
  Evaluation of the HIV reservoir size by measurement of 1) single copy HIV RNA quantification in samples with HIV RNA <50 copies/mL and 2) total HIV DNA and integrated HIV DNA in peripheral blood
Neuropsychological battery performance | Measured through week 96
  Evaluation of neuropsychological battery performance at week 48 and 96; and to later compare to RV 217 data from pre-infection and baseline early or acute HIV infection timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Polyak, MD, MPH, Study Chair — Henry M. Jackson Foundation in support of MHRP
Locations (1):
- Makerere University--Walter Reed Project (MUWRP), Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No